CLINICAL TRIAL: NCT00199576
Title: Prevention of Post-Extubation Laryngeal Edema With Intravenous Corticosteroids: a Prospective, Double-Blind, Placebo-Controlled Trial.
Brief Title: Prevention of Post-Extubation Laryngeal Edema With Intravenous Corticosteroids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AFSSAPS 001533; CIC0203/023
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Post-Extubation Laryngeal Edema
Keywords: Corticosteroids; Laryngotracheal injury; Intubation-extubation
MeSH Terms: interventions — Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone

SUMMARY:
Tracheal intubation is a frequent procedure in intensive care units (ICU). Post-extubation laryngeal edema is a frequent complication with potential morbidity and mortality, and may lead to urgent tracheal re-intubation. Corticosteroids have been proposed to reduce the incidence of post-extubation laryngeal edema. A few clinical studies have been conducted in adult ICU patients and have led to discrepant results. These discrepancies may be related to the time lag separating the administration of the corticosteroids and the planned extubation. Accordingly, we tested the hypothesis that pretreatment with corticosteroids initiated 12 hours before a planned extubation may efficiently prevent the occurrence of postextubation laryngeal edema in critically-ill adults who have been mechanically ventilated for more than 36 hours in the ICU.

DETAILED DESCRIPTION:
We conducted a prospective, double-blind, placebo-controlled, multicenter trial of 12-hour-pretreatment by methylprednisolone before a planned extubation in adult patients ventilated for more than 36 hours in the ICU. Methylprednisolone (20 mg) or placebo was first administered intravenously 12 hours before extubation and continued every 4 hours until tube removal. Primary endpoint was the occurrence of laryngeal edema within 24 hours of extubation. Laryngeal edema was clinically diagnosed and considered as major when requiring tracheal reintubation.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Intubated for ≥ 36 hours
* Scheduled extubation
* Informed written consent

Exclusion Criteria:

* pregnancy
* history of postextubation laryngeal dyspnea
* laryngeal disease
* tracheotomy
* patient receiving corticotherapy prior to admission
* traumatic intubation
* participation to this study or to another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670
Dates: Start 2000-12; Study Completion 2002-01

PRIMARY OUTCOMES:
Onset of a laryngeal edema within 24 hours after a planned tracheal extubation

SECONDARY OUTCOMES:
- Severity of laryngeal edema (minor or major)
- Time to onset of edema (in minutes) after tracheal extubation
- Need for a tracheal re-intubation

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bellissant, MD, PhD, Study Chair — CHU Rennes; Bruno Francois, MD, Principal Investigator — CH Limoges
Locations (15):
- France (15):
  - Réanimation médicale et chirurgicale - Hôpital d'Angoulême, Angoulême
  - Service de Réanimation - CH de Brive, Brivé
  - Service de Réanimation - CH de Chartres, Chartres
  - Service de Réanimation - CH de Chateauroux, Châteauroux
  - Réanimation polyvalente - Hôpital de Cholet, Cholet
  - Service de Réanimation - CH de Dreux, Dreux
  - Service de Réanimation - CH de Le Mans, Le Mans
  - Service de Réanimation Polyvalente - Hôpital Dupuytren, Limoges
  - Réanimation polyvalente - Hôpital d'Orléans, Orléans
  - Service Réanimation - CH de Poitiers, Poitiers
  - Service de Réanimation - CH de Saint Nazaire, Saint-Nazaire
  - Service de Réanimation - CH de Saintes, Saintes
  - Service de Réanimation - CH Saint Malo, St-Malo
  - Réanimation Médicale - Hôpital Bretonneau, Tours
  - Service de Réanimation - CH de Vannes, Vannes

REFERENCES:
- [Background] Kastanos N, Estopa Miro R, Marin Perez A, Xaubet Mir A, Agusti-Vidal A. Laryngotracheal injury due to endotracheal intubation: incidence, evolution, and predisposing factors. A prospective long-term study. Crit Care Med. 1983 May;11(5):362-7. doi: 10.1097/00003246-198305000-00009. PMID 6839788
- [Background] Darmon JY, Rauss A, Dreyfuss D, Bleichner G, Elkharrat D, Schlemmer B, Tenaillon A, Brun-Buisson C, Huet Y. Evaluation of risk factors for laryngeal edema after tracheal extubation in adults and its prevention by dexamethasone. A placebo-controlled, double-blind, multicenter study. Anesthesiology. 1992 Aug;77(2):245-51. doi: 10.1097/00000542-199208000-00004. PMID 1642342
- [Background] Ho LI, Harn HJ, Lien TC, Hu PY, Wang JH. Postextubation laryngeal edema in adults. Risk factor evaluation and prevention by hydrocortisone. Intensive Care Med. 1996 Sep;22(9):933-6. doi: 10.1007/BF02044118. PMID 8905428
- [Derived] Francois B, Bellissant E, Gissot V, Desachy A, Normand S, Boulain T, Brenet O, Preux PM, Vignon P; Association des Reanimateurs du Centre-Ouest (ARCO). 12-h pretreatment with methylprednisolone versus placebo for prevention of postextubation laryngeal oedema: a randomised double-blind trial. Lancet. 2007 Mar 31;369(9567):1083-9. doi: 10.1016/S0140-6736(07)60526-1. PMID 17398307